CLINICAL TRIAL: NCT02063919
Title: Association Between Confocal Laser Endomicroscopic (CLE) Features and Colorectal Mucosal Microbiome
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2014SDU-QILU-G01
Record Dates: First submitted 2014-01-29; First posted 2014-02-17 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Neoplasia; Colorectal Inflammation; Hyperplasia; Mucosal Microbiome
MeSH Terms: conditions — Hyperplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The mucosal metagenome was obtained from biopsy specimen.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- endomicroscopy
  Interventions: Other: the mucosal microbiome in the biopsy specimen was analysed

INTERVENTIONS:
Other: the mucosal microbiome in the biopsy specimen was analysed

SUMMARY:
The purpose of this study is to determine whether an association between endomicroscopic pattern and colorectal mucosal microbiome exists.

DETAILED DESCRIPTION:
The gut microbiome plays a pivotal role in the intestinal pathophysiology. The mucosal microbiome is in the front face of microbiome-host cross-talk. Confocal laser endomicroscopy (CLE) can provide realtime mucosal images during ongoing endoscopy. We hypothesized that the mucosal pattern, here evaluated by endomicroscopy, may constitute specific microbiome niches and participate the evolvement of the mucosal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age < 80 years old
* Scheduled for colonoscopy in Qilu Hospital

Exclusion Criteria:

* antibiotic usage within 2 months
* probiotic or prebiotic usage within 2 months
* ascites
* jaundice
* liver cirrhosis
* impaired renal function
* coagulopathy
* fever
* pregnancy
* breastfeeding
* inability to provide informed consent
* known allergy to fluorescein sodium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with indications for colonoscopy in Qilu Hospital outpatient and inpatient department are the study population of this study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The operational taxonomy unit in the colorectal mucosal microbiome. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD., MD., Principal Investigator — Department of gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China